CLINICAL TRIAL: NCT02114723
Title: Assessment of Mediacal Taping Concept Self-applied, in the Treatment of Primary Dysmenorrhea
Brief Title: Effectiveness of Medical Taping Concept in Primary Dysmenorrhea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Miguel Hernandez de Elche (Other)
Responsible Party: Principal Investigator, María Isabel Tomás-Rodríguez, PT, PT, MSC, Universidad Miguel Hernandez de Elche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: DPC-MITR-01-1
Record Dates: First submitted 2014-04-07; First posted 2014-04-15 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Primary Dysmenorrhea
Keywords: Mediacal Taping concept; Neuromuscular bandage; Physiotherapy techniques; Kinesio Tape
MeSH Terms: interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medical Taping Concept (Active Comparator): 3 band of a special and hypoallergenic tape, called Cure Tape ® (2 strips of 12 x 5 cm and 1 strip of 20 cm x 5 cm) are attached to the abdominal and lower back. One piece of 12 cm in length is applied right from below the navel and reached to where the pubic hair below, and another piece of 12 cm in length is applied to make a cross shape with the first piece (inside 11-12 dermatomes area). The piece of 20cm in length is placed horizontally to the lower back.
  The bandage is applied at the time that menstrual pain begins and is stuck to the skin for 4-5 days until menstrual pain disappears
  Interventions: Device: Medical Taping Concept
- Cross tape (Placebo Comparator): Two pieces of special and squared tape of 2.5 x 2 cm called Cross Tape ® are attached to the external side of the thigh at the hip joint area (outside 11-12 dermatomes area)
  Interventions: Device: Medical Taping Concept

INTERVENTIONS:
Device: Medical Taping Concept — The material used is a lengthways tape bandage of cotton with elastic properties, provided with a layer of anti-allergic adhesive in one of its sides that does not contain latex. This layer of glue is applied according to a special pattern so as to allow adequate transpiration.
  The bandage is applied at the time that menstrual pain begins and is stuck to the skin for 4-5 days until menstrual pain disappears
  Other Names: Cure Tape®; Kinesio Tape®; Kinesiotape Akraven; Kinesio® Tex; BB Tape (Bio balance tape); BB Lattice Tape

SUMMARY:
Determine the effectiveness of a proceeding under kinesio tape on pain and systemic symptoms most frequently described in primary dysmenorrhea.

DETAILED DESCRIPTION:
The aim of this study is to assess the analgesic efficacy of self-applied Medical Taping Concept in the treatment of primary dysmenorrhea .

To evaluate this effect, a total of 128 students from the University Miguel Hernández , with the following inclusion criteria, participated in this study: history of menstrual pain, aged between 18 and 39 years who have performed a gynecological check in the last 18 months and who have been diagnosed with any kind of primary dysmenorrhea.

A preliminary survey to identify valid students was made. Thereafter the participants were separated into two different groups (intervention group and placebo group) in order to request the completion of three questionnaires about the characteristics of menstrual pain and other demographic data for the next two menstrual cycles before the intervention. One survey included a graphic scale so the students could mark the start and the end of the symptoms associated with the menstrual cycle.

After that the principal researcher will interviewed with the participants to show them the correct auto-application of the menstrual bandage and placebo. Each students group will receive a triptych with information and pictures to the correct application of the adhesive strips.

Finally, during two new menstrual cycles, the participants will answer the same questionnaires to assess symptoms and menstrual pain while being worn adhesive strips (3 pieces of Kinesio tape - 20 cm x 5 cm Tape Cure ®-, applied to the abdominal and lower back, in the intervention group; 2 pieces of Cross Tape ® 2.5 cm x 2 cm -, in the hip joint, in the placebo group. Participants may do personal hygiene during the days of the menstrual cycle with their adhesives strips placed on oneself.

The size sample will be 128 girls. Differences will be contrasted in comparison of means (quantitative improvement, with an ANOVA) to evaluate the intervention. 18 girls were randomly chosen to obtain an estimation of the contrast parameters considered (means and standard variations). With this size sample and a significance of 5%, the investigators will have a power for the total sample for the contrasts of 80%.

To describe the variables, the investigators will use frequencies (absolute and relative) for the qualitative variables. For the quantitative variables, the investigators will use means plus standard variations.

To verify the homogeneity of the randomization the investigators will use tests based on the X2 (Pearson or Fisher) and t-test. The same procedure will be used to verify that the participants who quit the study have similar characteristics as those who remain.

The improvement will be analyzed quantitatively using ANOVA test. Dependent variable: pain after the intervention. Independent variables: pain before the intervention, changes in pharmacological therapy and intervention group. In the event of significant differences in the ANOVA models the investigators will use the Tukey post-hoc test, in order to determine where the differences exist between the two groups.

Qualitatively, the investigators will assess the improvement by calculating indicators of clinical relevance: relative risk (RR), absolute risk reduction (ARR), relative risk reduction (RRR), and number needed to treat (NNT).

All the analyses will be made at a significance of 5%. The confidence intervals (CI) will be calculated for the most relevant parameters. The analyses will be done using IBM SPSS Statistics 19.0.

ELIGIBILITY:
Inclusion Criteria:

* Women presenting menstrual pain grade 2-3 according to the classification of the severity of primary dysmenorrhea Andersch and Milsom.
* Have attended gynecological examination in the past 18 months and had ever diagnosed as having a gynecological disorder different from primary dysmenorrhea
* Not have been diagnosed with secondary dysmenorrhea
* Regular menstrual cycles (cycle typical range of 21 to 35 days)
* Do not use an intrauterine contraceptive device (IUD) or taking oral contraceptive pills
* Nulliparous

Exclusion Criteria:

* Women with mild dysmenorrhea (pain lower 4 in a numeric pain scale range 0-10);
* Women with irregular or infrequent menstrual cycles (outside the typical range of cycle 21 to 35 days);
* Women using an intrauterine contraceptive device (IUD) or taking oral contraceptive pills.
* Women who suffer from diseases diagnosed added
* Women to which it has undergone a surgical procedure for the treatment
* Provide skin lesions in the abdominal wall
* Use or abuse of drugs or alcohol
* Body mass index (BMI) between> 15.99 kg/m2 (maximum value of underweight according to WHO) and <25.00 kg m2 (maximum overweight according to WHO)

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 129 (Actual)
Dates: Start 2014-02; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Pain NRS (numeric rating scale) | Participants will be followed for 4 menstrual cycles, an expected average of 5 mounths
  Evaluations will be performed before, just after, 2 hours, 4 hours, 8 hours, 12 hours, 24 hours, and 48 hours after treatment. It will be measured in abdominal area, low back, lower limb and head.

SECONDARY OUTCOMES:
Number of analgesics requiring during menstruation | Participants will be followed for 4 menstrual cycles, an expected average of 5 mounths

OTHER OUTCOMES:
Quality of live | before/after intervention (5 mounths)
  Quality of live Questionnaire Euroquol-5D (EQ-5D)

CONTACTS AND LOCATIONS:
Overall Officials: María I Tomás-Rodríguez, PT, MSC, Principal Investigator — Universidad Miguel Hernández de Elche; José V Toledo-Marhuenda, PhD, Study Director — Universidad Miguel Hernández de Elche; Vicente F Gil-Guillén, MD, PhD, Study Director — Universidad Miguel Hernández de Elche; Antonio Palazón-Bru, MPH, Study Chair — Universidad Miguel Hernández de Elche
Locations (1):
- Universidad Miguel Hernández de Elche, Sant Joan d'Alacant, Alicante, Spain

REFERENCES:
- [Result] Lim C, Park Y, Bae Y. The effect of the kinesio taping and spiral taping on menstrual pain and premenstrual syndrome. J Phys Ther Sci. 2013 Jul;25(7):761-4. doi: 10.1589/jpts.25.761. Epub 2013 Aug 20. PMID 24259847
- [Result] Wefers c, Pijnappel H.F, Stolwijk N.M. Effect of Cure Tape® on menstrual pain in women with primary dysmenorrhea. Ned Tijdscr Fysiother 119(6): 193-197, 2009
- [Result] Garzón-Rodríguez, C. Analgessic effectiveness of Kinesio Taping versus abdominal massage in women with dysmenorrhea. Cuest. fisioter.42 (3): 302-311, 2013
- [Result] Akin M, Price W, Rodriguez G Jr, Erasala G, Hurley G, Smith RP. Continuous, low-level, topical heat wrap therapy as compared to acetaminophen for primary dysmenorrhea. J Reprod Med. 2004 Sep;49(9):739-45. PMID 15493566
- [Result] Dawood MY, Ramos J. Transcutaneous electrical nerve stimulation (TENS) for the treatment of primary dysmenorrhea: a randomized crossover comparison with placebo TENS and ibuprofen. Obstet Gynecol. 1990 Apr;75(4):656-60. PMID 2179780
- [Derived] Tomas-Rodriguez MI, Palazon-Bru A, Martinez-St John DRJ, Toledo-Marhuenda JV, Asensio-Garcia MDR, Gil-Guillen VF. Effectiveness of medical taping concept in primary dysmenorrhoea: a two-armed randomized trial. Sci Rep. 2015 Nov 13;5:16671. doi: 10.1038/srep16671. PMID 26564807
- See also: Kinesio Taping® Association International — http://www.kinesiotaping.com/